CLINICAL TRIAL: NCT01005394
Title: Acute Longitudinal Transcranial Magnetic Stimulation (TMS) After Stroke
Brief Title: Navigated Transcranial Magnetic Stimulation in Monitoring Stroke Recovery
Status: Terminated | Type: Observational
Why Stopped: Insufficient recruitment
Sponsor: Nexstim Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: DR-NE-002
Record Dates: First submitted 2009-10-30; First posted 2009-11-02 (Estimated); Last update posted 2015-04-16 (Estimated); Status verified 2015-04

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Navigated TMS: single arm study where all subjects will be studied using the Navigated TMS device
  Interventions: Device: Navigated TMS examination

INTERVENTIONS:
Device: Navigated TMS examination — diagnostic examination using a single pulse TMS paradigm to evaluate corticospinal motor tract integrity and its evolution after stroke
  Other Names: device: eXimia NBS system

SUMMARY:
The past 10 years of research in persons more than 6 months post stroke have shown certain types of rehabilitation can help "re-wire" the brain. Transcranial magnetic stimulation (TMS) can be used to monitor this re-wiring by mapping the brain's function (measuring brain activity). Recent research suggests that TMS can be used for both prognosis (determining future function) and to determine what type of rehabilitation therapy will work best after stroke. The purposes of this research study are to: 1) determine changes in brain activity during the first 6 months after stroke (to determine how the brain "re-wires"); 2) compare changes in recovery of motor function with changes in brain re-wiring; 3) determine the ability of TMS to "predict" functional outcome in the first 6 months after stroke.

The primary hypotheses are: 1) functional recovery will be correlated with TMS changes (as measure motor threshold (MT), motor evoked potentials (MEPs) and recruitment curves; 2) baseline TMS will predict future functional outcomes at 3 and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* one sided ischemic stroke confirmed by radiology
* 20-80 years old

Exclusion Criteria:

* hemorrhagic stroke
* brainstem stroke
* cerebellar stroke
* thalamic stroke
* seizure with the recent stroke
* any history of uncontrolled seizure
* history of epilepsy
* pregnancy or planning on getting pregnant during the next year
* MRI incompatibility (e.g. metal implants in body)
* recent history (past year) of alcohol and drug abuse (due to lack of follow up)

Other criteria include TMS exclusions: aneurysm clips, previous surgery over motor cortex, open craniotomy

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 20-80 years who have suffered a unilateral ischemic stroke and who will undergo motor rehabilitation at the study center will be asked to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2009-10; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
navigated transcranial magnetic stimulation examination and correlation with motor functional testing | Enrollment, week 2, week 4 , week 12 and week 24 post-stroke

SECONDARY OUTCOMES:
Safety of navigated transcranial magnetic stimulation examination | each examination

CONTACTS AND LOCATIONS:
Overall Officials: Kari Dunning, PhD,PT, Principal Investigator — University of Cincinnati
Locations (1):
- Drake Rehabilitation Center, Cincinnati, Ohio, United States